CLINICAL TRIAL: NCT06377735
Title: Bronchial Arterial Infusion Plus Bronchial Arterial Chemoembolization (BAI-BACE) for Advanced Lung Squamous Cell Carcinoma: a Multicenter Single-arm Phase II Study
Brief Title: BAI-BACE for Advanced Lung Squamous Cell Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhou Qunfang, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHEST-001
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Squamous Cell Carcinoma
Keywords: bronchial arterial infusion; bronchial arterial chemoembolization; paclitaxel; CalliSpheres; cis-platinum; advanced central squamous cell carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Intervention Model Description: Bronchial arterial infusion, bronchial arterial chemoembolization (BACE-BAI) procedure was performed as follows: Bronchial arteriography was performed to find tumor-feeding artery. After the catheter had been inserted into the tumor-feeding artery, paclitaxel (300 mg) was infused slowly at least 30 min. BAI (bronchial arterial infusion) chemotherapy was followed by BACE (Drug-eluting beads bronchial arterial chemoembolization); the CalliSpheres loaded with cis-platinum (30 mg) were infused into the tumor-feeding arteries until stasis or near-stasis of blood flow in the vessel was observed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BAI-BACE (Experimental): Bronchial arterial infusion, bronchial arterial chemoembolization (BACE-BAI)
  Interventions: Procedure: BAI-BACE

INTERVENTIONS:
Procedure: BAI-BACE — Bronchial arterial infusion, bronchial arterial chemoembolization (BACE-BAI) procedure was performed as follows: Bronchial arteriography was performed to find tumor-feeding artery. After the catheter had been inserted into the tumor-feeding artery, paclitaxel (300 mg) was infused slowly at least 30 min. BAI (bronchial arterial infusion) chemotherapy was followed by BACE (Drug-eluting beads bronchial arterial chemoembolization); the CalliSpheres loaded with cis-platinum (30 mg) were infused into the tumor-feeding arteries until stasis or near-stasis of blood flow in the vessel was observed.

SUMMARY:
Bronchial arterial infusion plus bronchial arterial chemoembolization (BAI-BACE) has been reported as non-first-line therapy to treat lung cancer in many hospitals in China. BAI, which uses chemotherapeutic drugs directly injected into the tumor and achieved a high concentration in a short time to kill the tumor. Then BACE could seal off the tumor vessels. In this study, we aim to describe the efficacy and safety of BAI-BACE as non-first-line for advanced lung squamous cell carcinoma.

DETAILED DESCRIPTION:
This study is a multicenter, interventional study to explore the efficacy, safety of BAI-BACE as non-first-line therapy for advanced central squamous cell carcinoma. Lung cancer is the leading cause of cancer-related death worldwide. Owing to the insidious symptom, most patients (about 75 %) are diagnosed at the advanced stage of the disease and, thus, cannot undergo resection. The central squamous cell carcinoma accounts for 25% of all cases of lung cancer. The first-line standard treatment for advanced central squamous cell carcinoma is combined chemoradiotherapy, and chemoradiotherapy is usually as the second-line. However, treatment failure is noted in many patients, and those patients often face the limited therapy choice and poor prognosis. Bronchial arterial infusion plus bronchial arterial chemoembolization (BAI-BACE) has been reported to treat lung cancer in many hospitals in China. BAI, which use chemotherapeutic drugs directly injected into the tumor and achieved a high concentration in a short time to kill the tumor. Then BACE could seal off the tumor vessels. The systemic toxicity of this surgery is low and tolerable. This study will provide clinical evidence that BACE-BAI will provide survival benefit for patients with advanced central squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Squamous cell carcinoma diagnosed by pathology, and central location by imaging;
2. Age 18-80;
3. Patients failed to the standard first-line or second-line treatment;
4. Tumors limited in the chest;
5. Tumors were fed by bronchial artery through CTA reconstruction;
6. Patents received PD-1 inhibitor or not were also included;
7. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-2;
8. Images within 2 weeks before inclusion;
9. Life expectancy more than 3 months;
10. Agreed to participated in this clinical trial;
11. Hemameba ≥3.0 x109/L, neutrophil ≥1.5x109/L, hemoglobin≥10.0 g/L, platelet≥100x 109/L, ALT; AST; bilirubin ≤1.5-fold normal, GFR≥60ml/min.

Exclusion Criteria:

1. Contraindication of BAI or BACE;
2. Under 18 years or over 75 years;
3. extra-chest metastases;
4. Receiving other antitumor treatment;
5. Severe infection or pregnancy;
6. Severe Pulmonary fibrosis and pulmonary artery;
7. liver, kidney or poor physical conditions;
8. Severe pleural effusion or pericardial effusion;
9. Life expectancy less than 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival (PFS) | 12 months
  Progression was defined as progressive disease by independent radiologic review

SECONDARY OUTCOMES:
Overall survival (OS) | 24 months
  OS is the length of time from the date of inclusion until death from any cause.
Objective response rate (ORR) | 12 months
  ORR, as determined based on tumor response according to RECIST 1.1, is defined as the proportion of all included patients whose best overall response (BOR) is either a complete response or partial response.
Adverse events | 24 months
  Safety will be evaluated according to the NCI CTCAE Version 4.03. All observations

CONTACTS AND LOCATIONS:
Overall Officials: Feng Duan, MD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General hospital, Beijing, Beijing Municipality, China